CLINICAL TRIAL: NCT02411461
Title: Early-onset Obesity and Cognitive Impairment in Children With Pseudohypoparathyroidism
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ashley Shoemaker, Assistant Professor of Pediatrics, Pediatric Endocrinology and Diabetes, Vanderbilt University Medical Center
Other Study IDs: VR7195; 1K23DK101689-01A1 (NIH)
Record Dates: First submitted 2015-02-25; First posted 2015-04-08 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Pseudohypoparathyroidism; Albright Hereditary Osteodystrophy
Keywords: Pediatric obesity; pseudohypoparathyroidism; Albright Hereditary Osteodystrophy
MeSH Terms: conditions — Pseudohypoparathyroidism; Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pseudohypoparathyroidism type 1a: Study group
- Healthy siblings: Control group
- Obese patients: Control group

SUMMARY:
Pseudohypoparathyroidism type 1a (PHP1a) is a rare disease that causes childhood obesity and learning difficulties. This study will investigate eating behaviors and perform cognitive testing on children with PHP1a. The investigators will compare their results to those of healthy siblings and other obese children.

DETAILED DESCRIPTION:
Pseudohypoparathyroidism type 1a (PHP1a) is a genetic disorder that causes early-onset, syndromic obesity and cognitive impairment. This study aims to evaluate eating behaviors, cognition and executive function in children with PHP1a, compared with healthy siblings and matched obese controls.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PHP1a, sibling of a patient with PHP1a or matched obese control

Exclusion Criteria (PHP1a):

* Treatment with appetite-altering drug or initiation of a new weight loss program in the past 3 months
* Type 2 diabetes

Exclusion Criteria (Controls):

* Obesity due to a genetic syndrome, growth hormone deficiency, untreated hypothyroidism, Cushing syndrome or exogenous glucocorticoid administration
* Weight loss greater than 10% over the previous 6 months
* Autism or other significant learning disorder
* Type 2 diabetes
* Other significant medical condition

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with pseudohypoparathyroidism type 1a (PHP1a), their healthy siblings and matched obese controls
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-12-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Shoemaker, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shoemaker AH, Lomenick JP, Saville BR, Wang W, Buchowski MS, Cone RD. Energy expenditure in obese children with pseudohypoparathyroidism type 1a. Int J Obes (Lond). 2013 Aug;37(8):1147-53. doi: 10.1038/ijo.2012.200. Epub 2012 Dec 11. PMID 23229731
- [Background] Wang L, Shoemaker AH. Eating behaviors in obese children with pseudohypoparathyroidism type 1a: a cross-sectional study. Int J Pediatr Endocrinol. 2014;2014(1):21. doi: 10.1186/1687-9856-2014-21. Epub 2014 Oct 15. PMID 25337124
- [Background] Landreth H, Malow BA, Shoemaker AH. Increased Prevalence of Sleep Apnea in Children with Pseudohypoparathyroidism Type 1a. Horm Res Paediatr. 2015;84(1):1-5. doi: 10.1159/000381452. Epub 2015 Apr 23. PMID 25925491
- [Background] Perez KM, Lee EB, Kahanda S, Duis J, Reyes M, Juppner H, Shoemaker AH. Cognitive and behavioral phenotype of children with pseudohypoparathyroidism type 1A. Am J Med Genet A. 2018 Feb;176(2):283-289. doi: 10.1002/ajmg.a.38534. Epub 2017 Nov 28. PMID 29193623
- See also: Vanderbilt PHP Research Group Website — http://www.facebook.com/pseudohypoparathyroidism

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pseudohypoparathyroidism Type 1a | Healthy Siblings | Obese Patients
Started | 16 | 8 | 15
Completed | 16 | 8 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pseudohypoparathyroidism Type 1a | Healthy Siblings | Obese Patients | Total
Number analyzed (Participants) | 16 | 8 | 15 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 8 | 15 | 39
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 11 | 26
  Male | 6 | 3 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 16 | 8 | 15 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intelligence Quotient
Description: Intelligence quotient as measured by Kaufman Brief Intelligence Test, 2nd Edition. This scale yields standard scores where the mean is 100 and one standard deviation is 15. Higher scores indicate better function.
Time Frame: one day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pseudohypoparathyroidism Type 1a | Healthy Siblings | Obese Patients
Number analyzed (Participants) | 16 | 8 | 15
units on a scale | 85.9 (17.2) | 104.3 (8.9) | 103.2 (11.5)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse events were recorded during the study visit only.
Arm/Group | Pseudohypoparathyroidism Type 1a | Healthy Siblings | Obese Patients
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No